CLINICAL TRIAL: NCT00257361
Title: D-Cycloserine Augmentation of Exposure and Response Prevention Treatment for Obsessive-Compulsive Disorder
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: PI left the university
Sponsor: University of Florida (Other)
Collaborators: Obsessive Compulsive Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None
Other Study IDs: IRB Protocol #639-2004; 00053428
Record Dates: First submitted 2005-11-18; First posted 2005-11-22 (Estimated); Last update posted 2013-09-30 (Estimated); Status verified 2011-08

CONDITIONS: Obsessive Compulsive Disorder
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Cycloserine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: D-Cycloserine

SUMMARY:
We propose to undertake an initial study of DCS to determine whether it has any short-term clinical benefits when added to standard ERP therapy in adults with OCD.

DETAILED DESCRIPTION:
Exposure and response prevention (ERP) has proven efficacy for OCD treatment in adults. Yet, ERP does not help all individuals, and those who benefit often remain somewhat symptomatic. Behavioral models for OCD treatment are based on two components. First, fears are acquired by the development of an association between a neutral stimulus and an aversive stimulus such the former acquires the aversive properties of the latter. The neutral stimulus is then designated as a conditioned stimulus (CS), and the original aversive stimulus is called an unconditioned stimulus (UCS). Second, the acquired fears can be unlearned through presentation of the CS in the absence of the UCS, a process known as extinction. On a neural level, ERP incorporates similar mechanisms to those involved in fear conditioning. Antagonists at the glutamatergic NMDA receptor, which is involved in learning and memory, block both fear learning and extinction. D-Cycloserine (DCS), a partial agonist at the N-methyl-D-aspartate (NMDA) glutamate receptor subtype, augments learning in animals and humans. Clinical application in animals and humans suggest that DCS facilitates the fear extinction process when taken prior to exposure to feared stimuli. An initial trial in acrophobic adults provided support for acute DCS dosing as facilitating extinction to fear. Given that ERP is based on extinction, it follows that DCS may augment ERP therapy providing enhanced treatment effects. With this in mind, we propose to undertake an initial study of DCS to determine whether it has any short-term clinical benefits when added to standard ERP therapy in adults with OCD.

ELIGIBILITY:
Inclusion Criteria:

1. a principal diagnosis of OCD assigned at pre-treatment, derived from the ADIS-IV, with a clinical severity rating of 4 or above;
2. 18-65 years of age; and,
3. an IQ of ³ 80.

Exclusion Criteria:

1. positive diagnosis of schizophrenia, other psychotic disorder, pervasive developmental disorder, organic brain syndrome, or mental retardation;
2. do not speak English;
3. are unwilling to attend twice weekly sessions; or,
4. is pregnant, breast feeding a child, or attempting to become pregnant (see below rationale)

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2005-07

PRIMARY OUTCOMES:
YBOCS

SECONDARY OUTCOMES:
Response rate

CONTACTS AND LOCATIONS:
Overall Officials: Eric Storch, Ph.D., Principal Investigator — University of Florida